CLINICAL TRIAL: NCT01351350
Title: A Phase I, Open Label, Dose Escalation Study of Oral Administration of MLN0128 in Combination With Paclitaxel, With/Without Trastuzumab, in Subjects With Advanced Solid Malignancies
Brief Title: Dose Escalation Study of MLN0128 in Combination With Paclitaxel, With/Without Trastuzumab, in Subjects With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INK128-003; U1111-1181-8192 (Other: WHO)
Record Dates: First submitted 2011-02-21; First posted 2011-05-10 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-06

CONDITIONS: Advanced Solid Malignancies; Hematologic Malignancies
Keywords: Solid tumor, mTORC1/2 inhibitors, HER2
MeSH Terms: conditions — Hematologic Neoplasms | interventions — sapanisertib; Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- MLN0128P 30 mg QW (Experimental): MLN0128 and paclitaxel (MLN0128P): MLN0128 30 mg, capsule, orally, once weekly (QW) + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase.
  Interventions: Drug: MLN0128; Drug: paclitaxel
- MLN0128P 40 mg QW (Experimental): MLN0128 40 mg, capsule, orally, once a week (QW) + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase.
  Interventions: Drug: MLN0128; Drug: paclitaxel
- MLN0128P 6 mg QD×3d QW (Experimental): MLN0128 6 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase.
  Interventions: Drug: MLN0128; Drug: paclitaxel
- MLN0128P 7 mg QD×3d QW (Experimental): MLN0128 7 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase.
  Interventions: Drug: MLN0128; Drug: paclitaxel
- MLN0128P 8 mg QD×3d QW (Experimental): MLN0128 8 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase.
  Interventions: Drug: MLN0128; Drug: paclitaxel
- MLN0128P 9 mg QD×3d QW (Experimental): MLN0128 9 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase.
  Interventions: Drug: MLN0128; Drug: paclitaxel
- MLN0128P 10 mg QD×3d QW (Experimental): MLN0128 10 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase.
  Interventions: Drug: MLN0128; Drug: paclitaxel
- MLN0128P 7 mg QD×5d QW (Experimental): MLN0128 7 mg, capsule, orally, once daily 5 days on/2 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase.
  Interventions: Drug: MLN0128; Drug: paclitaxel
- MLN0128P 8 mg QD×3d QW HER2- (Experimental): MLN0128 8 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in human epidermal growth factor receptor 2 negative (HER-) cancer participants until disease progression or unacceptable toxicity for up to 1 year in the Expansion Phase.
  Interventions: Drug: MLN0128; Drug: paclitaxel
- MLN0128PH 8 mg QD×3d QW HER2+ (Experimental): MLN0128 + paclitaxel + trastuzumab (MLN0128PH): MLN0128 8 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 plus trastuzumab 4 mg/kg loading dose on Day 1 followed by 2 mg/kg, intravenous each week of a 4-week cycle in HER+ cancer participants until disease progression or unacceptable toxicity for up to 1 year in the Expansion Phase.
  Interventions: Drug: MLN0128; Drug: paclitaxel; Drug: trastuzumab

INTERVENTIONS:
Drug: MLN0128 — MLN0128 capsules
Drug: paclitaxel — paclitaxel intravenous infusion
Drug: trastuzumab — trastuzumab intravenous infusion
  Arms: MLN0128PH 8 mg QD×3d QW HER2+

SUMMARY:
This is a Phase I, open label, dose escalation study of oral administration of MLN0128 in combination with paclitaxel, with/without trastuzumab, in participants with advanced solid malignancies.

DETAILED DESCRIPTION:
This is a Phase I, open-label study consisting of a dose escalation phase in advanced solid malignancies to determine the maximum tolerated dose (MTD) of oral administration of MLN0128 in 1 or more dosing schedules, combined with paclitaxel on Days 1, 8 and 15 of each cycle, followed by an expansion phase for further safety and preliminary efficacy.

Once the MTD is determined for each of the dosing schedules evaluated, a dose and schedule will be selected for the expansion phase, which may enroll participants into 2 arms in parallel:

* Arm A will consist of HER2- unknown cancer participants receiving MLN0128+paclitaxel
* Arm B will consist of HER2+ cancer participants receiving MLN0128+paclitaxel plus weekly trastuzumab

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written consent
* Locally advanced or metastatic solid tumors with the exception of primary brain tumor, and have failed or are not eligible for standard of care therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Ability to swallow oral medications
* For women of child-bearing potential, negative serum or urine pregnancy test within 14 days prior to the first study drug administration and use of physician-approved method of birth control from 30 days prior to 30 days following the last study drug administration
* Male participants must be surgically sterile or must agree to use physician-approved contraception during the study and for 30 days following the last study drug administration
* Clinical laboratory values as specified in the protocol
* For expansion phase (Arm A) - HER2-/unknown participants will be enrolled
* For expansion phase (Arm B) - HER2+ cancer participants will be enrolled

Exclusion Criteria:

* Diagnosis of primary brain tumor
* Have received prior cancer or other investigational therapy within 2 weeks prior to the first administration of study drug
* Known impaired cardiac function or clinically significant cardiac disease
* Known treatment with systemic corticosteroid within one week prior to the first administration of study drug
* Diabetes mellitus
* Human immunodeficiency virus (HIV) infection
* Known active cardiovascular disease condition as specified in protocol
* Pregnancy (positive serum or urine pregnancy test) or breast feeding
* Malabsorption due to prior gastrointestinal (GI) surgery, GI disease
* Other clinically significant co-morbidities

Please note that there are additional inclusion and exclusion criteria. The study center will determine if you meet all of the criteria.

Site personnel will explain the trial in detail and answer any question you may have if you do qualify for the study. You can then decide whether or not you wish to participate. If you do not qualify for the trial, site personnel will explain the reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-02-28 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Fort Myers, Florida
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Burris HA 3rd, Kurkjian CD, Hart L, Pant S, Murphy PB, Jones SF, Neuwirth R, Patel CG, Zohren F, Infante JR. TAK-228 (formerly MLN0128), an investigational dual TORC1/2 inhibitor plus paclitaxel, with/without trastuzumab, in patients with advanced solid malignancies. Cancer Chemother Pharmacol. 2017 Aug;80(2):261-273. doi: 10.1007/s00280-017-3343-4. Epub 2017 Jun 10. PMID 28601972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at three investigative sites in the United States from 28 February 2011 to 15 Sep 2017.
Pre-assignment Details: Participants with advanced solid malignancies enrolled in the dose escalation phase to establish MTD: MLN0128 6,7,8,9,10 mg QDx3d QW, 7mg QDx5d QW or 30, 40 mg QW. The expansion phase enrolled participants in either A: HER2- cancer participants, MLN0128 at MTD+paclitaxel or B: HER2+ cancer participants, MLN0128 at MTD+paclitaxel+trastuzumab.
Groups:
- MLN0128P 30 or 40 mg QW: MLN0128 and paclitaxel (MLN0128P): MLN0128 30 or 40 mg, capsule, orally, once weekly (QW) + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase until Maximum Tolerated Dose (MTD) was established (Up to 15.3 weeks).
- MLN0128P 6, 7, 8, 9 or 10 mg QD×3d QW: MLN0128 and paclitaxel (MLN0128P): MLN0128 6 , 7, 8, 9 or 10 mg, capsule, orally, once daily (QD) 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase until MTD was established (Up to 87.4 weeks).
- MLN0128P 7 mg QD×5d QW: MLN0128 and paclitaxel (MLN0128P): MLN0128 7 mg, capsule, orally, once daily 5 days on/2 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase until MTD was established (Up 65.4 weeks).
- Expansion Cohort MLN0128P 8 mg QD×3d QW HER2-: MLN0128 and paclitaxel (MLN0128P): MLN0128 8 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in human epidermal growth factor receptor 2 negative (HER-) cancer participants until disease progression or unacceptable toxicity for up to 1 year in the Expansion Phase (Up to 61.6 weeks).
- Expansion Cohort MLN0128PH 8mg QD×3d QW HER2+ Plus Trastuzumab: MLN0128 + paclitaxel + trastuzumab (MLN0128PH): MLN0128 8 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 plus trastuzumab 4 mg/kg loading dose on Day 1 followed by 2 mg/kg, intravenous each week of a 4-week cycle in HER+ cancer participants until disease progression or unacceptable toxicity for up to 1 year in the Expansion Phase (Up to 23.4 weeks).
Period: Overall Study
Arm/Group | MLN0128P 30 or 40 mg QW | MLN0128P 6, 7, 8, 9 or 10 mg QD×3d QW | MLN0128P 7 mg QD×5d QW | Expansion Cohort MLN0128P 8 mg QD×3d QW HER2- | Expansion Cohort MLN0128PH 8mg QD×3d QW HER2+ Plus Trastuzumab
Started (Here, started indicates the participants who were enrolled.) | 8 | 29 | 11 | 13 | 7
Treated | 8 | 29 | 10 | 13 | 7
Dose-escalation Evaluable | 7 | 23 | 10 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 29 | 11 | 13 | 7
Not completed — Disease Progression | 5 | 13 | 6 | 8 | 5
Not completed — Adverse Event | 1 | 10 | 1 | 2 | 0
Not completed — Participant Decision | 2 | 6 | 3 | 3 | 2
Not completed — Enrolled but not Treated | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Subjects as Treated (ASaT) population, which consisted of all enrolled participants who received at least 1 dose of MLN0128.
Groups:
- Expansion Cohort MLN0128PH 8mg QDx3d QW HER2+ Plus Trastuzumab: MLN0128 + paclitaxel + trastuzumab (MLN0128PH): MLN0128 8 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 plus trastuzumab 4 mg/kg loading dose on Day 1 followed by 2 mg/kg, intravenous each week of a 4-week cycle in HER+ cancer participants until disease progression or unacceptable toxicity for up to 1 year in the Expansion Phase (Up to 23.4 weeks).
- Total: Total of all reporting groups
Arm/Group | MLN0128P 30 or 40 mg QW | MLN0128P 6, 7, 8, 9 or 10 mg QD×3d QW | MLN0128P 7 mg QD×5d QW | Expansion Cohort MLN0128P 8 mg QD×3d QW HER2- | Expansion Cohort MLN0128PH 8mg QDx3d QW HER2+ Plus Trastuzumab | Total
Number analyzed (Participants) | 8 | 29 | 10 | 13 | 7 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (14.34) | 62.9 (9.57) | 58.1 (14.70) | 54.2 (14.46) | 58.1 (8.03) | 59.3 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 14 | 7 | 6 | 6 | 38
  Male | 3 | 15 | 3 | 7 | 1 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 8 | 28 | 10 | 12 | 6 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 1 | 0 | 2 | 0 | 3
  White | 8 | 27 | 10 | 10 | 7 | 62
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 29 | 10 | 13 | 7 | 67

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Phase: Maximum Tolerated Dose (MTD)
Description: MTD is the highest dose level at which the participants tolerate treatment without dose-limiting toxicities during the first cycle (28 days) of therapy.
Time Frame: Cycle 1: Days 1 to 28
Population: Safety Population included all participants who received at least one dose of study drug.
Measure: Number; unit: mg (QD×3d QW)
Groups:
- Dose Escalation: Participants from the Dose Escalation Phase who received at least 1 dose of study medication. MLN0128 6,7,8,9 or10 mg QD×3d QW, 30 or 40 mg QW, or 7 mg QD×5d QW of a 4-week cycle in combination with paclitaxel (80 mg/m^2) on Days 1, 8, and 15 of Cycle 1.
Arm/Group | Dose Escalation
Number analyzed (Participants) | 40
mg (QD×3d QW) | 8

2. Primary Outcome: Dose Escalation Phase: Number of Participants With at Least 1 Dose Limiting Toxicity (DLT)
Description: DLT was defined as any of the following occurring during Cycle 1 (Days 1-28) and attributable to MLN0128P: Grade ≥ 3 nonhematologic toxicity; Grade 3 thrombocytopenia with hemorrhage; Grade 4 neutropenia lasting > 7 days in the absence of growth factor support; Grade 4 neutropenia of any duration associated with fever 38.5 degrees C and/or infection; Any other Grade 4 hematologic toxicity; Inability to administer at least 75 % of doses of MLN0128 within Cycle 1 due to drug-related toxicity; Any clinically significant occurrence which the investigators and sponsor agree would place participants at undue safety risk; Participants who experienced an adverse event (AE) that met the definition for a DLT.
Time Frame: Cycle 1: Days 1 to 28
Population: Dose-Escalation evaluable population included participants who received ≥ 75% of planned doses of MLN0128 in Cycle 1 or stopped study drug before receiving 75% of doses because of study drug-related AEs (considered as DLT).
Measure: Number; unit: participants
Groups:
- MLN0128P 30 mg QW: MLN0128 30 mg, capsule, orally, once weekly (QW) + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase until MTD was established.
- MLN0128P 40 mg QW: MLN0128 40 mg, capsule, orally, once a week (QW) + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase until MTD was established.
- MLN0128P 6 mg QD×3d QW: MLN0128 6 mg, capsule, orally, once daily (QD) 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase until MTD was established.
- MLN0128P 7 mg QD×3d QW: MLN0128 7 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase until MTD was established.
- MLN0128P 8 mg QD×3d QW: MLN0128 8 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase until MTD was established.
- MLN0128P 9 mg QD×3d QW: MLN0128 9 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase until MTD was established.
- MLN0128P 10 mg QD×3d QW: MLN0128 10 mg, capsule, orally, once daily 3 days on/4 days off each week + paclitaxel 80 mg/m^2, 1 hour infusion, on Days 1, 8 and 15 of a 4-week cycle in the Dose Escalation Phase until MTD was established.
Arm/Group | MLN0128P 30 mg QW | MLN0128P 40 mg QW | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 8 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW | MLN0128P 7 mg QD×5d QW
Number analyzed (Participants) | 5 | 2 | 3 | 3 | 3 | 5 | 9 | 10
participants | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 2

3. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with Complete Response (CR) and Partial Response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Each cycle was a 28 day cycle. CR was defined as the disappearance of all target lesions and for non-target lesions, the disappearance of all non-target lesions and normalization of tumor marker level. PR was defined of at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD and for non-target lesions.
Time Frame: At screening and thereafter every 2 cycles of treatment until disease progression (Up to 65.8 weeks)
Population: Full Analysis Set (FAS) included all participants who received 1 or more doses of MLN0128 and have adequate baseline and post-baseline data collected.
Measure: Number; unit: percentage of participants
Arm/Group | MLN0128P 30 or 40 mg QW | MLN0128P 6, 7, 8, 9 or 10 mg QD×3d QW | MLN0128P 7 mg QD×5d QW | Expansion Cohort MLN0128P 8 mg QD×3d QW HER2- | Expansion Cohort MLN0128PH 8mg QDx3d QW HER2+ Plus Trastuzumab
Number analyzed (Participants) | 8 | 22 | 9 | 10 | 5
percentage of participants | 0 | 9 | 44 | 10 | 20

4. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for MLN0128
Description: Participants in the 6 mg QD×3d QW and 9 mg QD×3d QW were dosed with MLN0128 in conjunction with paclitaxel during Cycle 1 and Cycle 2 when PK was collected. Participants in the 7 mg QD×3d QW cohorts were dosed with paclitaxel during Cycle 1, but were subsequently switched to MLN0128 being dosed 24 hours after paclitaxel infusion Cycle 2 (i e, C2D2). In all the other dosing cohorts, MLN0128 was dosed 24 hours after paclitaxel infusion. Cycle 1: Data was collected at Day 1 for the 6, 7 and 9 mg QD×3d QW arms and at Day 2 for the 8 and 10 mg QD×3d QW, 7 mg QD×5d QW, 30 and 40 mg QW arms. Cycle 2: Data was collected at Day 1 for the 6 and 9 mg QD×3d QW arms and at Day 2 for the 7,8 and 10 mg QD×3d QW, 7 mg QD×5d QW, 30 and 40 mg QW arms.
Time Frame: Cycles 1 and 2: Day 1 or 2
Population: Pharmacokinetic (PK) population included all participants enrolled during Dose Escalation phase, received at least 1 dose of MLN0128 and had sufficient concentration-time data to calculate PK parameters, with data available for Cmax. Here, number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | MLN0128P 30 mg QW | MLN0128P 40 mg QW | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 8 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW | MLN0128P 7 mg QD×5d QW
Number analyzed (Participants) | 6 | 2 | 3 | 4 | 3 | 6 | 13 | 10
ng/mL
  Cycle 1 | 245.0 [136.00 to 456.00] | 345.5 [306.00 to 385.00] | 26.7 [19.10 to 40.30] | 31.1 [20.40 to 52.40] | 41.8 [19.80 to 79.70] | 34.2 [23.90 to 47.10] | 100.0 [57.50 to 162.00] | 53.5 [26.70 to 101.00]
  Cycle 2: number analyzed (Participants) | 5 | 1 | 3 | 2 | 3 | 3 | 8 | 6
  Cycle 2 | 242.2 [105.00 to 356.00] | 107.0 [107.00 to 107.00] | 33.8 [14.70 to 58.70] | 45.5 [40.40 to 50.50] | 53.1 [46.00 to 57.20] | 23.0 [10.80 to 36.60] | 80.1 [21.00 to 166.00] | 45.3 [11.60 to 79.50]

5. Secondary Outcome: Cmin: Minimum Observed Plasma Concentration for MLN0128
Description: as for outcome 4
Time Frame: Cycles 1 and 2: Day 1 or 2
Population: Due to the change in planned analysis, minimum plasma concentration data was not collected.
Arm/Group | MLN0128P 30 mg QW | MLN0128P 40 mg QW | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 8 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW | MLN0128P 7 mg QD×5d QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for MLN0128
Description: Participants in the 6 mg QD×3d QW and 9 mg QD×3d QW were dosed with MLN0128 in conjunction with paclitaxel during Cycle 1 and Cycle 2 when PK was collected. Participants in the 7 mg QD×3d QW cohorts were dosed with paclitaxel during Cycle 1, but were subsequently switched to MLN0128 being dosed 24 hours after paclitaxel infusion Cycle 2 (i.e., C2D2). In all the other dosing cohorts, MLN0128 was dosed 24 hours after paclitaxel infusion. Cycle 1: Data was collected at Day 1 for the 6, 7 and 9 mg QD×3d QW arms and at Day 2 for the 8 and 10 mg QD×3d QW, 7 mg QD×5d QW, 30 and 40 mg QW arms. Cycle 2: Data was collected at Day 1 for the 6 and 9 mg QD×3d QW arms and at Day 2 for the 7,8 and 10 mg QD×3d QW, 7 mg QD×5d QW, 30 and 40 mg QW arms.
Time Frame: Cycles 1 and 2: Day 1 or 2
Population: PK population included all participants enrolled during Dose Escalation phase, received at least 1 dose of MLN0128 and had sufficient concentration-time data to calculate PK parameters, with data available for Tmax. Here, number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Median (Full Range); unit: hours
Arm/Group | MLN0128P 30 mg QW | MLN0128P 40 mg QW | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 8 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW | MLN0128P 7 mg QD×5d QW
Number analyzed (Participants) | 6 | 2 | 3 | 4 | 3 | 6 | 13 | 10
hours
  Cycle 1 | 3.0 [0.50 to 5.92] | 3.0 [2.00 to 4.00] | 2.0 [2.00 to 3.83] | 3.0 [1.03 to 4.08] | 5.6 [1.02 to 5.65] | 4.1 [3.67 to 6.00] | 1.0 [0.53 to 2.17] | 1.6 [0.65 to 5.53]
  Cycle 2: number analyzed (Participants) | 5 | 1 | 3 | 2 | 3 | 3 | 8 | 6
  Cycle 2 | 2.0 [1.87 to 3.90] | 4.0 [4.00 to 4.00] | 4.0 [2.00 to 4.02] | 2.0 [1.97 to 2.00] | 1.0 [0.92 to 4.00] | 5.5 [2.00 to 6.00] | 2.0 [1.00 to 5.75] | 2.7 [0.50 to 5.72]

7. Secondary Outcome: Terminal Phase Elimination Half-life (T1/2) for MLN0128
Time Frame: Cycle 1 Day 1
Population: PK population consisted of all participants enrolled during the Dose Escalation phase of the study who received at least 1 dose of MLN0128 and had sufficient concentration-time data to calculate 1 or more PK parameters. T1/2 data is only available for 2 participants in the MLN0128P 6 mg QD×3d QW and 2 participants in the MLN0128P 7 mg QD×3d QW arm.
Measure: Mean (Full Range); unit: hours
Arm/Group | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW
Number analyzed (Participants) | 2 | 2
hours | 6.6 [6.36 to 6.91] | 7.2 [7.03 to 7.30]

8. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for MLN0128
Time Frame: Cycle 1 Day 1
Population: PK population consisted of all participants enrolled during the Dose Escalation phase of the study who received at least 1 dose of MLN0128 and had sufficient concentration-time data to calculate 1 or more PK parameters. AUC∞ data is only available for 2 participants in each the MLN0128P 6 mg QD×3d QW and MLN0128P 7 mg QD×3d QW arms.
Measure: Mean (Full Range); unit: ng*hr/mL
Arm/Group | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW
Number analyzed (Participants) | 2 | 2
ng*hr/mL | 206.5 [183.00 to 230.00] | 286.0 [269.00 to 303.00]

9. Secondary Outcome: AUC(0-6): Area Under the Plasma Concentration-time Curve From Time 0 to 6 Hours for MLN0128
Description: Participants in the 6 mg QD×3d QW and 9 mg QD×3d QW were dosed with MLN0128 in conjunction with paclitaxel during Cycle 1 and Cycle 2 when PK was collected. Participants in the 7 mg QD×3d QW cohorts were dosed with paclitaxel during Cycle 1, but were subsequently switched to MLN0128 being dosed 24 hours after paclitaxel infusion Cycle 2 (i e, C2D2). In all the other dosing cohorts, MLN0128 was dosed 24 hours after paclitaxel infusion. Cycle 1: Data was collected at Day 1 for the 6, 7 and 9 mg QD×3d QW arms and at Day 2 for the 8 and 10 mg QD×3d QW, 7 mg QD×5d QW, 30 and 40 mg QW arms. Cycle 2: Data was collected at Day 1 for the 6 and 9 mg QD×3d QW arms and at Day 2 for the 7,8 and 10 mg QD×3d QW, 30 and 40 mg QW arms.
Time Frame: Cycles 1 and 2: Day 1 or 2
Population: PK population included all participants enrolled during Dose Escalation phase, received at least 1 dose of MLN0128 and had sufficient concentration-time data to calculate PK parameters. Here, number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Full Range); unit: ng*hr/mL
Arm/Group | MLN0128P 30 mg QW | MLN0128P 40 mg QW | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 8 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW
Number analyzed (Participants) | 6 | 2 | 3 | 4 | 3 | 6 | 13
ng*hr/mL
  Cycle 1 | 753.7 [428.00 to 1290.00] | 1325.0 [1210.00 to 1440.00] | 104.4 [73.70 to 146.00] | 121.7 [82.70 to 187.00] | 139.9 [58.00 to 282.00] | 146.2 [99.20 to 229.00] | 347.0 [203.00 to 505.00]
  Cycle 2: number analyzed (Participants) | 5 | 1 | 3 | 2 | 3 | 3 | 8
  Cycle 2 | 883.6 [464.00 to 1340.00] | 505.0 [505.00 to 505.00] | 106.8 [55.50 to 165.00] | 174.0 [162.00 to 186.00] | 210.3 [143.00 to 253.00] | 72.6 [28.10 to 144.00] | 283.9 [65.60 to 660.00]

10. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Paclitaxel
Time Frame: Cycles 1 and 2: Day 1
Population: PK population included all participants enrolled during Dose Escalation phase, received at least 1 dose of paclitaxel and had sufficient concentration-time data to calculate PK parameters, with data available for Cmax. Here, number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | MLN0128P 30 mg QW | MLN0128P 40 mg QW | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 8 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW | MLN0128P 7 mg QD×5d QW
Number analyzed (Participants) | 5 | 2 | 3 | 4 | 3 | 6 | 13 | 10
ng/mL
  Cycle 1, Day 1 | 2538.0 [1090.00 to 3220.00] | 2355.0 [2210.00 to 2500.00] | 1933.3 [1280.00 to 3170.00] | 1942.5 [1540.00 to 2420.00] | 1620.0 [1290.00 to 1990.00] | 3798.3 [1270.00 to 11100.00] | 2906.9 [2090.00 to 4020.00] | 1637.7 [410.00 to 2770.00]
  Cycle 2, Day 1: number analyzed (Participants) | 4 | 1 | 3 | 2 | 3 | 3 | 5 | 6
  Cycle 2, Day 1 | 3462.5 [2300.00 to 4210.00] | 1500.0 [1500.00 to 1500.00] | 1200.3 [421.00 to 2090.00] | 1550.0 [1550.00 to 1550.00] | 3103.3 [1440.00 to 4890.00] | 1602.3 [597.00 to 2350.00] | 2964.0 [1560.00 to 4070.00] | 1765.7 [654.00 to 2670.00]

11. Secondary Outcome: Cmin: Minimum Observed Plasma Concentration for Paclitaxel
Description: as for outcome 4
Time Frame: Cycles 1 and 2: Day 1 or 2
Population: Due to the change in planned analysis, minimum plasma concentration data was not collected.
Arm/Group | MLN0128P 30 mg QW | MLN0128P 40 mg QW | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 8 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW | MLN0128P 7 mg QD×5d QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Paclitaxel
Time Frame: Cycles 1 and 2: Day 1
Population: PK population consisted of all participants enrolled during Dose Escalation phase of study who received at least 1 dose of MLN0128 or paclitaxel and had sufficient concentration-time data to calculate PK parameters for either compound. Here, number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Median (Full Range); unit: hours
Arm/Group | MLN0128P 30 mg QW | MLN0128P 40 mg QW | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 8 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW | MLN0128P 7 mg QD×5d QW
Number analyzed (Participants) | 5 | 2 | 3 | 4 | 3 | 6 | 13 | 10
hours
  Cycle 1, Day 1 | 1.1 [1.02 to 1.17] | 1.1 [1.03 to 1.17] | 1.1 [1.00 to 1.15] | 1.2 [0.87 to 1.55] | 1.2 [1.08 to 1.62] | 1.1 [1.00 to 2.22] | 1.1 [0.52 to 1.87] | 1.5 [1.00 to 1.88]
  Cycle 2, Day 1: number analyzed (Participants) | 4 | 1 | 3 | 2 | 3 | 3 | 5 | 6
  Cycle 2, Day 1 | 1.1 [1.00 to 1.47] | 1.2 [1.2 to 1.2] | 1.6 [1.0 to 1.6] | 1.4 [1.20 to 1.50] | 1.2 [1.07 to 1.75] | 1.2 [1.08 to 1.83] | 1.0 [0.95 to 1.17] | 1.1 [1.02 to 1.55]

13. Secondary Outcome: Terminal Phase Elimination Half-life (T1/2) for Paclitaxel
Time Frame: Cycle 1 Day 1
Population: PK population consisted of all participants enrolled during the Dose Escalation phase of the study who received at least 1 dose of paclitaxel and had sufficient concentration-time data to calculate 1 or more PK parameters. T1/2 data is only available for participants in the MLN0128P 6,7,9 and 10 mg QD×3d QW arms.
Measure: Mean (Full Range); unit: hours
Arm/Group | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW
Number analyzed (Participants) | 2 | 3 | 5 | 2
hours | 10.0 [9.93 to 10.00] | 9.1 [8.83 to 9.48] | 9.6 [8.19 to 11.60] | 9.3 [9.10 to 9.53]

14. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Paclitaxel
Time Frame: Cycle 1 Day 1
Population: PK population consisted of all participants enrolled during the Dose Escalation phase of the study who received at least 1 dose of paclitaxel and had sufficient concentration-time data to calculate 1 or more PK parameters. AUC∞ data is only available for participants in the MLN0128P 6,7,9 and 10 mg QD×3d QW arms.
Measure: Mean (Full Range); unit: ng*hr/mL
Arm/Group | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW
Number analyzed (Participants) | 2 | 3 | 5 | 2
ng*hr/mL | 4590.0 [3440.00 to 5740.00] | 4790.0 [4040.00 to 6270.00] | 5002.0 [2910.00 to 6330.00] | 5485.0 [4550.00 to 6420.00]

15. Secondary Outcome: AUC(0-6): Area Under the Plasma Concentration-time Curve From Time 0 to 6 Hours for Paclitaxel
Time Frame: Cycle 1 Day 1
Population: Participants from the PK population, all participants enrolled during the Dose Escalation phase of the study who received at least 1 dose of paclitaxel and had sufficient concentration-time data to calculate 1 or more PK parameters, with data available for analyses.
Measure: Mean (Full Range); unit: ng*hr/mL
Arm/Group | MLN0128P 30 mg QW | MLN0128P 40 mg QW | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 8 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW | MLN0128P 7 mg QD×5d QW
Number analyzed (Participants) | 6 | 2 | 3 | 4 | 3 | 6 | 13 | 10
ng*hr/mL | 3198.3 [1560.00 to 4140.00] | 3515.0 [2930.00 to 4100.00] | 2620.0 [1800.00 to 3970.00] | 3157.5 [2810.00 to 3550.00] | 2683.3 [1820.00 to 3630.00] | 5315.0 [1880.00 to 15100.00] | 3683.8 [2600.00 to 5330.00] | 2657.0 [1140.00 to 5350.00]

16. Secondary Outcome: AUC(0-24): Area Under the Plasma Concentration-time Curve Extrapolated to 24 Hours for Paclitaxel
Time Frame: Cycle 1 Day 1
Population: PK population consisted of all participants enrolled during the Dose Escalation phase of the study who received at least 1 dose of paclitaxel and had sufficient concentration-time data to calculate 1 or more PK parameters. AUC0-24 data is only available for participants in the MLN0128P 6,7,9 and 10 mg QD×3d QW arms.
Measure: Mean (Full Range); unit: ng*hr/mL
Arm/Group | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW
Number analyzed (Participants) | 3 | 4 | 6 | 2
ng*hr/mL | 3583.3 [2510.00 to 5160.00] | 4332.5 [3670.00 to 5510.00] | 6415.0 [2550.00 to 15900.00] | 5135.0 [4290.00 to 5980.00]

17. Secondary Outcome: CL: Total Clearance Calculated Using the Observed Value of the Last Quantifiable Concentration for Paclitaxel
Time Frame: Cycle 1 Day 1
Population: PK population consisted of all participants enrolled during the Dose Escalation phase of the study who received at least 1 dose of paclitaxel and had sufficient concentration-time data to calculate 1 or more PK parameters. CL data is only available for participants in the MLN0128P 6,7,9 and 10 mg QD×3d QW arms.
Measure: Mean (Full Range); unit: L/hr
Arm/Group | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW
Number analyzed (Participants) | 2 | 3 | 5 | 2
L/hr | 36.2 [24.70 to 47.70] | 34.8 [22.30 to 45.30] | 31.2 [22.30 to 48.20] | 25.8 [19.30 to 32.30]

18. Secondary Outcome: Vss: Volume of Distribution at Steady State Calculated Using the Observed Value of the Last Quantifiable Concentration for Paclitaxel
Time Frame: Cycle 1 Day 1
Population: PK population consisted of all participants enrolled during the Dose Escalation phase of the study who received at least 1 dose of paclitaxel and had sufficient concentration-time data to calculate 1 or more PK parameters. Vss data is only available for participants in the MLN0128P 6,7,9 and 10 mg QD×3d QW arms.
Measure: Mean (Full Range); unit: L
Arm/Group | MLN0128P 6 mg QD×3d QW | MLN0128P 7 mg QD×3d QW | MLN0128P 9 mg QD×3d QW | MLN0128P 10 mg QD×3d QW
Number analyzed (Participants) | 2 | 3 | 5 | 2
L | 313.5 [189.00 to 438.00] | 262.0 [219.00 to 306.00] | 252.2 [149.00 to 441.00] | 150.0 [120.00 to 180.00]

19. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs), Serious Adverse Events(SAEs), AEs Resulting in Discontinuation of MLN0128 and Fatal AEs Within 30 Days of Last Dose of Study Drug
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A serious adverse event is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: First dose of study drug through 30 days after the administration of the last dose of study drug (Up to approximately 91.4 weeks)
Population: All Subjects as Treated (ASaT) population consisted of all enrolled participants who received at least 1 dose of MLN0128, was used in the safety analyses.
Measure: Number; unit: percentage of participants
Arm/Group | MLN0128P 30 or 40 mg QW | MLN0128P 6, 7, 8, 9 or 10 mg QD×3d QW | MLN0128P 7 mg QD×5d QW | Expansion Cohort MLN0128P 8 mg QD×3d QW HER2- | Expansion Cohort MLN0128PH 8mg QDx3d QW HER2+ Plus Trastuzumab
Number analyzed (Participants) | 8 | 29 | 10 | 13 | 7
percentage of participants
  TEAE | 100 | 100 | 100 | 100 | 100
  SAE | 63 | 41 | 60 | 31 | 43
  Fatal AEs within 30 Days of Last Dose Study Drug | 25 | 7 | 20 | 15 | 14
  AEs Resulting in Discontinuation of MLN0128 | 13 | 34 | 10 | 15 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug through 30 days after the administration of the last dose of study drug (Up to approximately 91.4 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. According to the protocol analysis planned, data was collected as per the dosing schedule.
Arm/Group | MLN0128P 30 or 40 mg QW | MLN0128P 6, 7, 8, 9 or 10 mg QD×3d QW | MLN0128P 7 mg QD×5d QW | Expansion Cohort MLN0128P 8 mg QD×3d QW HER2- | Expansion Cohort MLN0128PH 8mg QD×3d QW HER2+ Plus Trastuzumab
All-Cause Mortality (participants affected / at risk) | 2/8 | 2/29 | 2/10 | 2/13 | 1/7
Serious Adverse Events (participants affected / at risk) | 5/8 | 12/29 | 6/10 | 4/13 | 3/7
Other Adverse Events (participants affected / at risk) | 8/8 | 29/29 | 10/10 | 13/13 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN0128P 30 or 40 mg QW (N=8) | MLN0128P 6, 7, 8, 9 or 10 mg QD×3d QW (N=29) | MLN0128P 7 mg QD×5d QW (N=10) | Expansion Cohort MLN0128P 8 mg QD×3d QW HER2- (N=13) | Expansion Cohort MLN0128PH 8mg QD×3d QW HER2+ Plus Trastuzumab (N=7)
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 2 | 2 | 0 — One treatment-emergent death occurred during treatment with 8 mg QDx3d QW HER2- dose cohort and is not related.
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with 40 mg MLN0128 QW dose cohort and is not related.
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 — Two treatment-emergent death occurred during treatment with 40 mg QW and 9 mg MLN0128 QD×3d QW dose cohort and are not related.
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with MLN0128 8 mg QD×3d QW HER2+ Plus Trastuzumab dose cohort and is not related.
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with 8 mg QDx3d QW HER2- dose cohort and is not related.
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Tracheal obstruction extrinsic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with 7 mg MLN0128 QD×5d QW dose cohort and is not related
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Disease Progression (General disorders) | 0 | 1 | 0 | 0 | 0 — Two treatment-emergent death occurred during treatment with 9 mg MLN0128 QD×3d QW and 7 mg QD×5d QW dose cohort and are not related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MLN0128P 30 or 40 mg QW (N=8) | MLN0128P 6, 7, 8, 9 or 10 mg QD×3d QW (N=29) | MLN0128P 7 mg QD×5d QW (N=10) | Expansion Cohort MLN0128P 8 mg QD×3d QW HER2- (N=13) | Expansion Cohort MLN0128PH 8mg QD×3d QW HER2+ Plus Trastuzumab (N=7)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 14 | 3 | 3 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 8 | 3 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 12 | 7 | 4 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 7 | 3 | 1 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 18 | 6 | 6 | 6
Constipation (Gastrointestinal disorders) | 3 | 4 | 2 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 5 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 3
Gastritis (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 12 | 3 | 4 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 3 | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pharyngeal lesion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4 | 3 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 3 | 5 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 2 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 4 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Nail bed tenderness (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 11 | 4 | 4 | 2
Pyrexia (General disorders) | 2 | 4 | 0 | 3 | 1
Oedema peripheral (General disorders) | 0 | 3 | 2 | 2 | 1
Chills (General disorders) | 1 | 2 | 1 | 0 | 1
Pain (General disorders) | 0 | 2 | 2 | 2 | 0
Feeling jittery (General disorders) | 0 | 0 | 0 | 1 | 0
Puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 7 | 1 | 4 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 5 | 0 | 3 | 2
Dysgeusia (Nervous system disorders) | 0 | 4 | 1 | 2 | 1
Headache (Nervous system disorders) | 1 | 4 | 1 | 3 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 1 | 5 | 1
Syncope (Nervous system disorders) | 0 | 2 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 2 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 2 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 2 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 2 | 6 | 0 | 5 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 3 | 1 | 1
Low density lipoprotein increased (Investigations) | 0 | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 1 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 2 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0
High density lipoprotein decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Protein total decreased (Investigations) | 1 | 0 | 0 | 2 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood cholosterol increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1
Carbon dioxide increased (Investigations) | 0 | 0 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 4 | 2 | 0 | 0
Hypotension (Vascular disorders) | 1 | 4 | 1 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 4 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 2 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 1 | 0 | 1
Visual impairment (Eye disorders) | 1 | 1 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 1 | 0
Orbital Oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Arhropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 2 | 2 | 2
Claustrophobia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 2
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 15 | 6 | 7 | 4
Vomiting (Gastrointestinal disorders) | 5 | 10 | 3 | 7 | 6
Stomatitis (Gastrointestinal disorders) | 2 | 13 | 4 | 5 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 12 | 2 | 3 | 1
Fatigue (General disorders) | 4 | 19 | 8 | 9 | 4
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 2 | 0
Peripheral swelling (General disorders) | 0 | 1 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 8 | 4 | 3 | 0
Urinary tract infection (Infections and infestations) | 3 | 5 | 4 | 4 | 2
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Paranasal Sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 3 | 0 | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 4 | 1 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Superior vena cava occlusion (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Burn oral cavity (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2013-10-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT01351350/SAP_000.pdf
  • Study Protocol (2014-03-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT01351350/Prot_001.pdf